CLINICAL TRIAL: NCT01717170
Title: Study of the Safety, Tolerability, and Bioactivity of Tocilizumab On Patients With Non-infectious UVEITIS: The STOP-UVEITIS Study
Acronym: STOP-Uveitis
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Nebraska (Other)
Responsible Party: Principal Investigator, Quan Dong Nguyen, MD, Professor and Chair, University of Nebraska
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ML28522
Record Dates: First submitted 2012-10-26; First posted 2012-10-30 (Estimated); Last update posted 2017-04-28 (Actual); Status verified 2017-04

CONDITIONS: Intermediate Uveitis; Posterior Uveitis; Pan-uveitis
Keywords: Non-infectious Uveitis, Tocilizumab
MeSH Terms: conditions — Uveitis, Intermediate; Uveitis, Posterior | interventions — tocilizumab

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tocilizumab (4 mg/kg) (Experimental): Tocilizumab (4 mg/kg) as an intravenous infusion over 1 hour at day 0, 30, 60, 90, 120, and 150.
  Interventions: Drug: Tocilizumab
- Tocilizumab (8 mg/kg) (Experimental): Tocilizumab (8 mg/kg) as an intravenous infusion over 1 hour at day 0, 30, 60, 90, 120, and 150.
  Interventions: Drug: Tocilizumab

INTERVENTIONS:
Drug: Tocilizumab — Tocilizumab (4 mg/kg or 8 mg/kg)
  Other Names: ACTEMRA

SUMMARY:
In the STOP-UVEITIS study, we propose to evaluate the safety, tolerability, and bioactivity of two doses of Tocilizumab (4mg/kg and 8mg/kg), administered monthly, in patients with non-infectious intermediate, posterior, or panuveitis.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18;
* Able to give informed consent and attend all study visits;
* Have diagnosis of uveitis determined by the Investigator to be non-infectious;
* Have active uveitis, defined as having at least 1+ Vitreous Haze (SUN scale) in study eye. As mentioned above, at least 12 of the randomized subjects must also have vitreous haze of ≥ 2+ vitreous haze. and:
* are receiving no other treatment; or,
* are receiving prednisone ≥10 mg/day (or equivalent dose of another corticosteroid) and/or at least 1 other systemic immunosuppressant;
* Have posterior, intermediate, or panuveitis; for panuveitis, if an anterior component is present, it must be less than the posterior component;
* Sufficient inflammation to require systemic treatment or long-term regional treatment. Patients whom the investigators feel may only need short-term topical therapy should not be enrolled.
* Best-corrected EARLY TREATMENT DIABETIC RETINOPATHY STUDY(ETDRS) visual acuity of 20/20 to 20/400 (approximately 80 to 20 letters) in the study eye;
* Best- corrected ETDRS visual acuity of 20/400 or better in the fellow eye (approximately 20 letters).
* Must have a chest radiograph within 3 months prior to enrollment with no evidence of malignancy, infection or fibrosis.
* Females of childbearing potential must have a negative serum pregnancy test at screening. In addition, sexually active females of childbearing potential must agree to use TWO of the following adequate forms of contraception while on study medication: oral, injectable, or implantable hormonal contraceptives; tubal ligation; intrauterine device; barrier contraceptive with spermicide; or vasectomized partner.
* Males must agree to use barrier contraception (latex condoms) when engaging in sexual activity while on study medication and for 28 days after taking the last dose of study medication.
* Subjects with a documented history of non-infectious intermediate-, anterior and intermediate, posterior, or pan-uveitis including but not restricted to: intermediate uveitis, sarcoidosis, Vogt-Koyanagi-Harada (VKH) syndrome, birdshot retinochoroidopathy, retinal vasculitis, sympathetic ophthalmia, multifocal choroiditis with panuveitis. Prior to study screening, potential subjects must have been evaluated and screened for infectious etiologies by the investigators, possibly as part of standard clinical acre; all testing to rule out infectious causes must be performed within 3 months of screening for the STOP-UVEITIS study.
* Currently active and uncontrolled uveitis (of the types mentioned above) that at the determination of the investigator, requires the initiation of corticosteroid monotherapy at a dose of ≥ 10 mg/day (or equivalent) or prednisone therapy and immunomodulatory therapy or injections of corticosteroid (intravitreal or periocular); or uveitis in subjects for whom oral corticosteroid is contraindicated, relatively or absolutely.
* Evidence of active non-infectious ocular inflammation, that at the determination of investigator, requires therapy (e.g. vitreous cells, vitreous haze, retinal vasculitis, chorioretinitis). Such evidence can be documented by clinical examination, photography, or ancillary testing (e.g. fluorescein angiography, indocyanine green (ICG), optical coherence tomography). As long as the investigator determines that the degree of inflammation can be monitored for regression or progression, the inflammation criterion can be met.
* Not planning to undergo elective ocular surgery during the first 6 months of the study.

Exclusion Criteria:

* Any significant ocular disease that could compromise vision in the study eye. These include, but are not limited to:

  * Diabetic retinopathy: proliferative diabetic retinopathy (PDR) or non-proliferative diabetic retinopathy (NPDR) that compromise the vision.
  * Age-related macular degeneration;
  * Myopic degeneration with active subfoveal choroidal neovascularization.
  * Advanced glaucoma status post trabeculectomy or tube/valve placement
* Any of the following treatments within 90 days prior to Day 0 or anticipated use of any of the following treatments to the study eye:

  * Intravitreal injections (including but not limited to steroids or anti-vascular endothelial growth factors);
  * Posterior subtenon's steroids
* Intraocular surgery within 90 days prior to Day 0 in the study eye;
* Capsulotomy within 30 days prior to Day 0 in the study eye;
* History of vitreoretinal surgery or scleral buckling
* Any ocular surgery (including cataract extraction or capsulotomy) of the study eye anticipated within the first 180 days following Day 0;
* Intraocular pressure (IOP) ≥25 mmHg in the study eye (glaucoma patients maintained on no more than 2 topical medications with IOP <25 mmHg are allowed to participate);
* Pupillary dilation inadequate for quality stereoscopic fundus photography in the study eye;
* Media opacity that would limit clinical visualization;
* Presence of any form of ocular malignancy in the study eye, including choroidal melanoma;
* History of herpetic infection in the study eye or adnexa;
* Presence of known active or inactive toxoplasmosis in either eye;
* Ocular or periocular infection in either eye;
* Participation in other investigational drug or device clinical trials within 30 days prior to Day 0, or planning to participate in other investigational drug or device clinical trials within 180 days following Day 0. This includes both ocular and non-ocular clinical trials
* Major surgery (including joint surgery) within 8 weeks prior to screening or planned major surgery within 6 months following randomization
* Prior treatment with any cell-depleting therapies, including investigational agents or approved therapies, some examples are CAMPATH, anti-CD4, anti-CD5, anti¬CD3, anti-CD19 and anti-CD20
* Treatment with intravenous gamma globulin, plasmapheresis or Prosorba column within 6 months of baseline
* Immunization with a live/attenuated vaccine within 4 weeks prior to baseline
* Previous treatment with tocilizumab (TCZ)
* Any previous treatment with alkylating agents such as chlorambucil, or with total lymphoid irradiation
* History of severe allergic or anaphylactic reactions to human, humanized or murine monoclonal antibodies
* Evidence of serious uncontrolled concomitant cardiovascular, nervous system, pulmonary (including obstructive pulmonary disease), renal, hepatic, endocrine (include uncontrolled diabetes mellitus) or gastrointestinal disease (including complicated diverticulitis, ulcerative colitis, or Crohn"s disease)
* Current liver disease as determined by principal investigator unless related to primary disease under investigation
* Known active current or history of recurrent bacterial, viral, fungal, mycobacterial or other infections (including but not limited to tuberculosis and atypical mycobacterial disease, Hepatitis B and C, and herpes zoster, but excluding fungal infections of nail beds)
* Any major episode of infection requiring hospitalization or treatment with IV antibiotics within 4 weeks of screening or oral antibiotics within 2 weeks prior to screening
* Active tuberculosis (TB) requiring treatment within the previous 3 years. Patients should be screened for latent TB and, if positive, treated following local practice guidelines prior to initiating (Tocilizumab)TCZ. Patients treated for tuberculosis with no recurrence in 3 years are permitted
* Primary or secondary immunodeficiency (history of or currently active)
* Evidence of active malignant disease, malignancies diagnosed within the previous 5 years (including hematological malignancies and solid tumors, except basal and squamous cell carcinoma of the skin or carcinoma in situ of the cervix uteri that has been excised and cured)
* Pregnant women or nursing (breast feeding) mothers
* Patients with reproductive potential not willing to use an effective method of contraception
* History of alcohol, drug or chemical abuse within 1 year prior to screening.
* Neuropathies or other conditions that might interfere with pain evaluation unless related to primary disease under investigation
* Patients with lack of peripheral venous access
* Serum creatinine > 1.6 mg/dL (141 μmol/L) in female patients and > 1.9 mg/dL(168 μmol/L) in male patients. Patients with serum creatinine values exceeding limits may be eligible for the study if their estimated glomerular filtration rates (GFR) are >30.
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 1.5 times upper limit of normal (ULN)
* Total Bilirubin > ULN
* Platelet count < 100 x 109/L (100,000/mm3)
* Hemoglobin < 85 g/L (8.5 g/dL; 5.3 mmol/L)
* White Blood Cells < 3.0 x 109/L (3000/mm3)
* Absolute Neutrophil Count < 2.0 x 109/L (2000/mm3)
* Absolute Lymphocyte Count < 0.5 x 109/L (500/mm3)
* Positive Hepatitis BsAg, or Hepatitis C antibody

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2013-03; Primary Completion 2017-06 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Frequency and severity of adverse events from baseline (BL) to month 6. | Baseline (BL) to month 6.
  Safety and tolerability of repeated Tocilizumab infusions in patients with non-infectious uveitis, as assessed by frequency and severity of adverse events from baseline (BL) to month 6.

SECONDARY OUTCOMES:
Frequency and severity of adverse events at month 12. | Baseline to Month 12
  Safety and tolerability of repeated Tocilizumab infusions in patients with non-infectious uveitis, as assessed by frequency and severity of adverse events at month 12.

OTHER OUTCOMES:
Percentage of patients with a decrease of ≥ 2 steps in vitreous haze or resolution of haze (for patients with 1+ haze at baseline) based on the National Eye Institute (NEI) scale at 1, 3, 6, and 12 months after therapy or at time of rescue. | Months 1, 3, 6, and 12 after therapy or at the time of rescue therapy administration.
  Percentage of patients with a decrease of ≥ 2 steps in vitreous haze or resolution of haze (for patients with 1+ haze at baseline) based on the National Eye Institute (NEI) scale at 1, 3, 6, and 12 months after therapy or at time of rescue. All patients who receive rescue therapy will be followed until the conclusion of month 12.

CONTACTS AND LOCATIONS:
Overall Officials: Quan D Nguyen, MD, MSc, Principal Investigator — Truhlsen Eye Institute, University of Nebraska Medical Center
Locations (1):
- Truhlsen Eye Institute, University Of Nebraska Medical Center, Omaha, Nebraska, United States

REFERENCES:
- [Derived] Sadiq MA, Hassan M, Afridi R, Halim MS, Do DV, Sepah YJ, Nguyen QD; STOP-UVEITIS Investigators. Posterior segment inflammatory outcomes assessed using fluorescein angiography in the STOP-UVEITIS study. Int J Retina Vitreous. 2020 Oct 6;6:47. doi: 10.1186/s40942-020-00245-w. eCollection 2020. PMID 33042579